CLINICAL TRIAL: NCT04663906
Title: Does Oral Isotretinoin Increase the Risk of Developing Infection With and Complications From Covid-19, Compared to an Age-matched Background Population
Brief Title: Oral Isotretinoin and Covid-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 1/095/20
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Isotretinoin Adverse Reaction; Covid19
Keywords: isotretinoin; Covid19; coronavirus; covid-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isotretinoin: Test population, prescribed oral isotretinoin between March and October 2020.
- Control: Background age-matched population, not prescribed oral isotretinoin during March to October 2020

SUMMARY:
There is a theoretical risk that the nasal mucosal dryness caused by oral retinoid medications may increase the risk of patients becoming infected with Covid-19.

Isotretinoin is a drug used commonly in dermatology, usually for management of acne and occasionally for management of other dermatological diseases. The most common side effect of oral isotretinoin is mucocutaneous dryness, which can lead to nasal dryness and crusting. Isotretinoin is derived from vitamin A and produces this side effect by arresting the cell cycle of mucus secreting cells in the nasal cavity. The mucus usually secreted moisturises the nasal cavity and provides a protective, lubricating layer overlying the cilia.

Cilia and nasal mucous are both believed to have roles in defence against infection and immunity. Hence it was postulated at the start of the pandemic that the effect this medication has on the nasal environment may increase the likelihood of contracting a disease spread by droplet or aerosol particles.

In March 2020 we established a departmental Excel database of our patients on oral retinoid medications in order to track those currently receiving treatment.

The database includes people taking isotretinoin, alitretinoin and acitretin. The greatest number of patients in this database are in the isotretinoin group and patients taking isotretinoin tend to be a relatively young and fit population. Acitretin on the other hand is often used in an older population who may have other underlying disease comorbidities. There were only a very small number of patients taking alitretinoin in the database.

In order to limit confounding variables and provide as clear a result as possible, it was decided to limit this study to comparing the group of patients taking isotretinoin, aged 16-40years, with an age-matched background population from NHS Grampian.

This study would examine the electronic patient record of patients aged 16-40years, taking isotretinoin between March and October 2020 and compare their rates of Covid-19 infection, hospitalisation and complications with the rates of the local age-matched background population. Persons taking isotretinoin in the time period would be excluded from the background population.

As Covid-19 is a new disease, the existing research literature on this specific topic is extremely limited, and so far this study would be the first in this area.

DETAILED DESCRIPTION:
Isotretinoin is a drug used commonly in dermatology, usually for management of acne and occasionally for management of other dermatological diseases. The most common side effect of oral isotretinoin is mucocutaneous dryness, which can lead to nasal dryness and crusting. Isotretinoin is derived from vitamin A and produces this side effect by arresting the cell cycle of mucus secreting cells in the nasal cavity. The mucus usually secreted moisturises the nasal cavity and provides a protective, lubricating layer overlying the cilia.

Cilia and nasal mucous are both believed to have roles in defence against infection and immunity. Hence it was postulated at the start of the pandemic that the effect this medication has on the nasal environment may increase the likelihood of contracting a disease spread by droplet or aerosol particles, such as Covid-19.

In March 2020 we established a departmental database of our patients on oral retinoid medications in order to track those currently receiving treatment. The database includes people taking isotretinoin, alitretinoin and acitretin. The greatest number of patients in this database are in the isotretinoin group and patients taking isotretinoin tend to be a relatively young and fit population. Acitretin on the other hand is often used in an older population who may have other underlying disease comorbidities. There were only a very small number of patients taking alitretinoin in the database.

In order to limit confounding variables and provide as clear a result as possible, it was decided to limit this study to comparing the group of patients taking isotretinoin, aged 16-40years, with an age-matched background population from NHS Grampian.

This study would examine the electronic patient record of patients aged 16-40years, taking isotretinoin between March and October 2020 and compare their rates of Covid-19 infection, hospitalisation and complications with the rates of the local age-matched background population. Persons taking isotretinoin in the time period would be excluded from the background population.

As Covid-19 is a new disease, the existing research literature on this specific topic is extremely limited, and so far this study would be the first in this area.

The electronic patient record of patients aged 16-40years taking isotretinoin between March and October 2020 will be accessed and the following will be recorded:

* Covid-19 testing while on or within 4 weeks after treatment
* Positive Covid-19 test while on or within 4 weeks after treatment
* Hospitalisation with Covid-19 while on or within 4 weeks after treatment
* ICU admission while on or within 4 weeks of treatment
* Death directly attributed to Covid-19 while on or within 4 weeks of treatment. The data held in the database is identifiable and held on the NHS Grampian secure server.

Once the details above are filled in each case will be anonymised with a case number. A key linking this back to the CHI will be kept on the NHS Grampian secure server.

Further data analysis will be completed using the anonymised data.

Details of an age matched local population can be obtained from Health Intelligence pending R&D approval of this study.

The University of Aberdeen department of medical statistics have already been consulted about this project and are willing to offer their help with data analysis. Once statistical analysis has been decided upon we will update the protocol or submit the details as an amendment, before analysis takes place.

ELIGIBILITY:
Inclusion Criteria:

* Test: prescribed oral isotretinoin in NHS Grampian age 16-40years includive, between March-Oct 2020

Background control population: residing in NHS Grampian, age 16-40years, etsted for Covid-19 between march -oct 2020, not prescribed oral isotretinoin in timeframe.

Exclusion Criteria:

* Test population: not prescribed oral isotretinoin in NHS grampian, outwith age range 16-40years or treatment range March-October 2020.

Background control popuat8ion: prescribed oral isotretinoin between march-october 2020, age outwith 16-40years, not tested for covid-19 between March-Oct 2020.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This is an estimate based on the number of patients taking isotretinoin aged 16-40 we have in the departmental database. We would try and obtain equal numbers in the isotretinoin and background populations as far as possible, roughly 125 patients who received isotretinoin and 125 background patients who did not. The numbers in each population can only be finally determined when the database is interrogated and details are obtained from Health Intelligence, neither of which can happen prior to approvals
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | March - October 2020
  Did patients taking isotretinoin have a greater risk of infection with Covid-19 compared to an age-matched background population not taking isotretinoin.

SECONDARY OUTCOMES:
Secondary Outcome | March - October 2020
  Did patients taking isotretinoin have a greater risk of hospitalisation related to Covid-19, ICU admission, or death from Covid-19, compared to an age-matched background population not taking isotretinoin

IPD SHARING:
Plan to Share IPD: No
Patient data will be reviewed bu study team only.